CLINICAL TRIAL: NCT00077779
Title: A Multi-Center Randomized, Double-Blind, Placebo-Controlled Study of the Human Anti-TNF Monoclonal Antibody Adalimumab for the Induction and Maintenance of Clinical Remission in Subjects With Crohn's Disease
Brief Title: Adalimumab for the Induction and Maintenance of Clinical Remission in Subjects With Crohn's Disease
Acronym: CHARM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M02-404
Record Dates: First submitted 2004-02-12; First posted 2004-02-16 (Estimated); Last update posted 2007-09-26 (Estimated); Status verified 2007-09

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Adalimumab

INTERVENTIONS:
Drug: Adalimumab

SUMMARY:
The purpose of this study is to test whether Adalimumab (at two different doses) can induce and maintain clinical remission in subjects with active Crohn's disease when compared to placebo (a substance containing no medication)

ELIGIBILITY:
Inclusion:

* Males and females between the ages of 18 and 75 who are diagnosed with moderate to severe Crohn's Disease defined by a CDAI score of >= 220 and <= 450, normal laboratory parameters,
* are willing and able to give informed consent, and
* are able to self-inject or have a designee or healthcare professional who can inject the study medication.

Exclusion:

* History of certain types of cancer, diagnosis of ulcerative colitis,
* female or breast feeding subjects,
* surgical bowel resection(s) with in the past 6 months,
* history of listeria,
* human immunodeficiency virus (HIV),
* central nervous system demyelinating disease or untreated TB,
* history of a poorly controlled medical condition,
* unsuccessful response to infliximab or any anti-TNF agent use in the past.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 854 (Actual)
Dates: Start 2003-07

PRIMARY OUTCOMES:
Clinical remission (CDAI<150). | 56 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul F Pollack, M.D., Study Director — Abbott
Locations (43):
- United States (43):
  - Thornton Hospital Reumatology Division, La Jolla, California
  - UCSF San Francisco General Hospital, San Francisco, California
  - Cal-West, Inc., San Francisco, California
  - Western States Clinical Research, Arvada, Colorado
  - Gastroenterology Associates of Fairfield County, Bridgeport, Connecticut
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - V.A. Medical Center, Gainsville, Florida
  - Mark Lamet, MD, Hollywood, Florida
  - Gastroenterology Consultants, Ormond Beach, Florida
  - Northwest Gastroenterology, Arlington Heights, Illinois
  - Northwestern University, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - Indianapolis Gastroenterology Research Foundation, Indianapolis, Indiana
  - St. Vincent Hospital: Research Department, Indianapolis, Indiana
  - Drug Research Services, Inc., Metairie, Louisiana
  - Maryland Clinical Trials, Annapolis, Maryland
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Capital Gastroenterology Consultants, P.A., Silver Spring, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Mayo Clinic Research, Rochester, Minnesota
  - Gastroenterology & Hematology, Kansas City, Missouri
  - Glenn Gordon, MD, Mexico, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Washington University School, St Louis, Missouri
  - Long Island Clinical Research Assoc., Great Neck, New York
  - NY Center for Clinical Research, Lake Success, New York
  - Daniel Present, MD, New York, New York
  - Digestive Disease Associates of Rockland, Pomona, New York
  - Charlotte Gastroenterology & Hepatology, Charlotte, North Carolina
  - Carolina Digestive Health Associates, Charlotte, North Carolina
  - Carolina Research Associates, Charlotte, North Carolina
  - Le Bauer Research, P.A., Greensboro, North Carolina
  - Wilmington Gastroenterology, Wilmington, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Westhills Gastroenterology, Portland, Oregon
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Columbia Gastro Associates, Columbia, South Carolina
  - Gastroenterology Center of the Mid South, Memphis, Tennessee
  - Nashville Medical Research, Nashville, Tennessee
  - Gastrointestinal Specialists, Richmond, Virginia
  - Discovery Research Inteternational, LLC, Milwaukee, Wisconsin
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Sandborn WJ, Lewis JD, Panes J, Loftus EV, D'Haens G, Yu Z, Huang B, Lacerda AP, Pangan AL, Feagan BG. Association Between Proposed Definitions of Clinical Remission/Response and Well-Being in Patients With Crohn's Disease. J Crohns Colitis. 2022 Mar 14;16(3):444-451. doi: 10.1093/ecco-jcc/jjab161. PMID 34546360
- [Derived] Ryan C, Sobell JM, Leonardi CL, Lynde CW, Karunaratne M, Valdecantos WC, Hendrickson BA. Safety of Adalimumab Dosed Every Week and Every Other Week: Focus on Patients with Hidradenitis Suppurativa or Psoriasis. Am J Clin Dermatol. 2018 Jun;19(3):437-447. doi: 10.1007/s40257-017-0341-6. PMID 29380251
- [Derived] Panaccione R, Colombel JF, Sandborn WJ, D'Haens G, Zhou Q, Pollack PF, Thakkar RB, Robinson AM. Adalimumab maintains remission of Crohn's disease after up to 4 years of treatment: data from CHARM and ADHERE. Aliment Pharmacol Ther. 2013 Nov;38(10):1236-47. doi: 10.1111/apt.12499. Epub 2013 Sep 22. PMID 24134498
- [Derived] Schreiber S, Reinisch W, Colombel JF, Sandborn WJ, Hommes DW, Robinson AM, Huang B, Lomax KG, Pollack PF. Subgroup analysis of the placebo-controlled CHARM trial: increased remission rates through 3 years for adalimumab-treated patients with early Crohn's disease. J Crohns Colitis. 2013 Apr;7(3):213-21. doi: 10.1016/j.crohns.2012.05.015. Epub 2012 Jun 16. PMID 22704916
- [Derived] Kamm MA, Hanauer SB, Panaccione R, Colombel JF, Sandborn WJ, Pollack PF, Zhou Q, Robinson AM. Adalimumab sustains steroid-free remission after 3 years of therapy for Crohn's disease. Aliment Pharmacol Ther. 2011 Aug;34(3):306-17. doi: 10.1111/j.1365-2036.2011.04717.x. Epub 2011 Jun 5. PMID 21645018
- [Derived] Colombel JF, Schwartz DA, Sandborn WJ, Kamm MA, D'Haens G, Rutgeerts P, Enns R, Panaccione R, Schreiber S, Li J, Kent JD, Lomax KG, Pollack PF. Adalimumab for the treatment of fistulas in patients with Crohn's disease. Gut. 2009 Jul;58(7):940-8. doi: 10.1136/gut.2008.159251. Epub 2009 Feb 6. PMID 19201775